CLINICAL TRIAL: NCT04026646
Title: The Effects of Proprioceptive Neuromuscular Facilitation and Static Stretching Exercises on Proprioceptive Sensation and Performance
Brief Title: The Effects of Proprioceptive Neuromuscular Facilitation and Static Stretching Exercises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/09-13
Record Dates: First submitted 2019-07-03; First posted 2019-07-19 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Flexibility
Keywords: Flexibility; Proprioception; Physical Performance
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation stretching exercises (Experimental): Proprioceptive Neuromuscular Facilitation stretching exercises (contract-relax-antagonist-contract method) will be performed 6 repetition and totally 30 seconds stretching for hamstring muscle group will be performed.
  Interventions: Procedure: Proprioceptive Neuromuscular Facilitation stretching exercise
- Static stretching exercises (Experimental): Passive Static Stretching exercises will be performed 2 repetition and totally 30 seconds stretching for hamstring muscle group will be performed.
  Interventions: Procedure: Static stretching exercise

INTERVENTIONS:
Procedure: Proprioceptive Neuromuscular Facilitation stretching exercise — Proprioceptive Neuromuscular Facilitation stretching exercises (contract-relax-antagonist-contract method) will be performed 6 repetition and totally 30 seconds stretching for hamstring muscle group will be performed.It will be applied 3 days in a week for 8 week.
  Arms: Proprioceptive Neuromuscular Facilitation stretching exercises
Procedure: Static stretching exercise — Static stretching exercises will be applied 2 repetition. Totally 30 seconds stretching for hamstring muscle group will be performed. It will be applied 3 days in a week for 8 week.
  Arms: Static stretching exercises

SUMMARY:
In this randomized trial, the aim of study is compare acute and chronic effect of Proprioceptive Neuromuscular Facilitation stretching and static stretching in individuals with shortness hamstring in proprioception and performance. The primary outcome measurement is proprioception (position sense and motion sense), the secondary outcome measurements are physical performance evaluations.

All exercises will be performed by the same physiotherapist in 8 weeks and 3 times a week. Exercises will be performed bilaterally and data from the dominant lower extremity will be used in the analysis. Exercises and assessments to reduce the effects of circadian variation will be performed at the same times during the research.

DETAILED DESCRIPTION:
Joint proprioception can be defined as the body's ability to determine position and detection movement without vision perception. Proprioception is provided from the stimulation of specialized nerve endings and mechanoreceptors located in and around the joints, such as muscles, tendons, fascia, joint capsule, and ligaments. The muscle spindle and golgi tendon organ are the most important receptors involved in the proprioceptive sensation of the knee joint.

In the literature, there are studies have investigated the effect of static stretching exercises on the sense of position. Some of these studies showed an improvement on position sense, while one study showed no effect. There are a limited number of studies have investigated the effects of Proprioceptive Neuromuscular Facilitation (PNF) stretching techniques on proprioceptive senses. However, the effects of static stretching and PNF stretching on kinesthesia have not been studied.

The aim of this study is to compare acute and chronic effect of PNF stretching and static stretching in individuals with shortness hamstring in proprioception and performance.

Hypothesis of research

H01: The acute effects of static stretching and PNF stretching exercises on the results of proprioceptive sensation are similar.

H02: The chronic effects of static stretching and PNF stretching exercises on the results of proprioceptive sensation are similar.

H03: The acute effects of static stretching and PNF stretching exercises on the results of physical performance are similar.

H04: The chronic effects of static stretching and PNF stretching exercises on the results of physical performance are similar.

The Universe and Sample of the Research:

A sample size calculation was performed using the G* Power software (version 3.1.9.2), taking into account the statistical tests to be used in the analyses, and the conventional effect size values proposed by Cohen. It was estimated that 27 subjects would be needed in each group (α=0.05, β=0.20, and Cohen d=0.8) in order to detect statistically significant difference in a Mann Whitney U test. Considering the samples that could not complete the study, this first sample size was increased by 10% and the final sample size was calculated as 30 in each group.

Methods:

The study will include volunteer sedentary male subjects aged between 20-29 years. The study will be carried out in the athlete's lab of the Eastern Mediterranean University.

Participants in the study who have signed a voluntary consent form will be informed about the study. Then, the evaluation starts with the socio-demographic data of the participants (age, gender, height, weight, dominant side). Evaluations will be performed as knee extension angle, proprioceptive sense, flexibility assessment, balance, explosive power tests and muscle strength assessment. Individuals will be divided into two groups by minimization randomization method. 30 seconds contract-relax-antagonist-contract method (CRAC) of Proprioceptive Neuromuscular Facilitation stretching exercises for hamstring muscle will be performed to Group 1 and 30 seconds static stretching exercises for hamstring muscle will be performed to Group 2.

To assess the acute effect, exercise will be performed after the first assessment and then all assessments will be repeated. To investigate the chronic effect, all exercises will be performed in 8 weeks and 3 times a week. After 6 weeks follow-up period, all participants will be evaluated again.

Evaluations in the Research

Knee Extension Test:

The individual's hip will be stabilized at 90 degrees flexion with 1 hand supporting the subject's distal thigh and the other hand cupping the heel. Physiotherapist passively extended the knee until the individual feels mild tension in hamstring muscle. At this point, it will measured the angle using a goniometer. Full knee extension would be equivalent to an angle of 180°. The angle missing from the full knee extension will be recorded as 'degree'.

Proprioceptive Sensory Measurements:

Isokinetic dynamometer will be used to evaluate the knee joint proprioceptive sense of subjects. The subjects will placed in a 90° hip flexion sitting position. Subjects will be informed about the tests. Before the test, a trial will be performed. Between the three tests 30 seconds rest period will be given. The difference between the target angle and the measured angle will be registered as absolute error. Averages of three measurements will be analyzed.

For motion sense measurements, 10° knee flexion position was selected for kinesthesia measurements. The subjects will be instructed to press the dynamometer lock button as soon as they will perceive any movement in the knee joint. 45° knee flexion position will be used in the measurement of position sense. The knee will be started in the 90° flexion position and before the test, target knee position will be taught during 5 seconds. Afterwards, the knee will be placed to starting position. Subjects will be asked to push the warning button as soon as they feel they will reach the target angle.

Room temperature will be kept at 25°C during the tests. Air splints will be used to eliminate the tactile sense. While care will be taken to preserve the silence of the environment, subjects will be dressed in headphones at the same time to prevent the sound coming from the isokinetic dynamo-meter that will affect the measurements.

Flexibility Measurement:

It will be evaluated using the sit and reach test. Individuals will be asked to reach the as far as possible they can reach by extending their arms to the forward and stand still for 1-2 seconds at the last point without bending participants' knees. The distance will be recorded in 'cm' and the best value will be used in the analysis.

Balance Measurements:

Flamingo Balance Test:

Static balance will be measured by Flamingo Balance Test. The subjects stood on the beam which was 50 cm long, 5 cm height and 3 cm wide. While balancing on the dominant leg, the free leg was flexed at the knee and the foot of this leg held close to the buttocks. Then the instructor will be started the stopwatch and the subjects tried to stand in this position for one minute. The stopwatch will be stopped each time the subjects lost the balance during 60 second. The number of falls of the individual will be recorded. The test will be repeated 3 times and a rest interval of 60 seconds will be given between repetitions. The best result will be recorded.

Y-Balance Test:

Dynamic balance will be measured with Y-balance test. Individuals will be asked to place one foot on the starting point on the center and both hands on the waist. Individuals will be reach the farthest point possible in the anterior, posteriomedial and posteriolateral directions with the free limb. The farthest point of the free limb will be measured with the tape measure. There will be 3 trials in each direction. In addition, the lower extremity length measurement will be used for scoring. (Spina Iliaca Anterior Superior-Medial Malleoli). The mixed reach distance will be calculated based on best value [(max anterior + max posteriomedial + max posteriolateral) / (3 x Lower Limb Length)] x100.

Anaerobic Power Tests:

Vertical Jump Test:

Explosive force of lower extremities will be evaluated using the counter movement vertical jump test. The tape measure will be placed and fixed on the wall in the vertical direction. The individuals will be positioned on the side of the wall. In this position, the arm will be extended and the point at which the longest finger reaches will be recorded. The subject will be started with their hands on their hips, they will then instructed to sink (approximately 120 knee angle) as high as possible. The distance between the touched point and jumped points on the tape measure will be measured and recorded in 'cm'. The test will be repeated 3 times and a rest interval of 60 seconds will be given between repetitions. The best result will be recorded.

Horizontal Jump Test:

Explosive force of lower extremities will be evaluated using the counter movement horizontal jump test. The tape measure will be placed horizontally and fixed on the hard ground. The individuals will be positioned on the '0' point of the tape measure. In this position, the arm will be extended and the point at which the longest finger reaches will be recorded. The subject will be jump with their hands on their hips (approximately 120 knee angle) as forward as possible with the double leg. The distance between the '0' point and jumped points on the tape measure will be measured and recorded in 'cm'. The test will be repeated 3 times and a rest interval of 60 seconds will be given between repetitions. The best result will be recorded.

Muscle Strength:

The evaluation of quadriceps and hamstring muscle concentric strength will be evaluated with the isokinetic dynamometer. Before the measurements, the bike will be used for warming for 5 minutes without resistance. The test will be performed 5 times at 120 ̊/sec angular speeds. The peak torque values of the results will be recorded in 'N / m'.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-29 years of age,
* Male individuals,
* Individuals who have not participated in physical activity for the last 6 months,
* Who have the knee extension angle more than 20⁰,
* Who accept the conditions of the study and sign the written informed consent form.

Exclusion Criteria:

* Patients who have lower extremity injuries in the last 6 months,
* Who have visual or vestibular impairments except of refractive problems,
* Who have traumatic problems, who have rheumatologic, orthopedic or neuromuscular disease, Black people (due to muscle structure).

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-03-08 (Estimated)

PRIMARY OUTCOMES:
Change between baseline of Knee Extension test and after 8th week | The test will be performed 2 times. Assessment will be performed baseline and after 8th weeks. Measurement takes about 5 minutes.
  The knee extension test will be evaluated with goniometer.
Change between baseline of Position Sense test and after 8th week | The test will be performed 2 times. Assessment will be performed baseline and after 8th weeks. Measurement takes about 5 minutes.
  The position sense will be evaluated with isokinetic dynamometer.
Change between baseline of Motion Sense and after 8th week | The test will be performed 2 times. Assessment will be performed baseline and after 8th weeks. Measurement takes about 5 minutes.
  The motion sense will be evaluated with isokinetic dynamometer.

SECONDARY OUTCOMES:
Change between baseline of Knee Extension Test and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 5 minutes.
  The knee extension test will be evaluated with goniometer.
Change on Knee Extension Test after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 5 minutes.
  The knee extension test will be evaluated with goniometer.
Change between baseline of Position Sense test and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 5 minutes.
  The position sense will be evaluated with isokinetic dynamometer.
Change on Position Sense test after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 5 minutes.
  The position sense will be evaluated with isokinetic dynamometer.
Change between baseline of Motion Sense test and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 5 minutes.
  The motion sense will be evaluated with isokinetic dynamometer.
Change on Motion Sense after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 5 minutes.
  The motion sense will be evaluated with isokinetic dynamometer.
Change between baseline of Flexibility and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 5 minutes.
  Flexibility will be evaluated by the sit-reach test in cm.
Change between baseline of Flexibility and after 8th week | Assessment will be performed baseline and after 8th weeks. Measurement takes about 5 minutes.
  Flexibility will be evaluated by the sit-reach test in cm.
Change on Flexibility after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 5 minutes.
  Flexibility will be evaluated by the sit-reach test in cm.
Change between baseline of Static Balance and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 5 minutes.
  Static balance will be evaluated by the Flamingo Balance Test.
Change between baseline of Static Balance and after 8th week stretching exercise | Assessment will be performed baseline and after 8th weeks. Measurement takes about 5 minutes.
  Static balance will be evaluated by the Flamingo Balance Test.
Change on Static Balance after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 5 minutes.
  Static balance will be evaluated by the Flamingo Balance Test.
Change between baseline of Dynamic Balance and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 10 minutes.
  Static balance will be evaluated by the Y Balance Test.
Change between baseline of Dynamic Balance and after 8th week stretching exercise | Assessment will be performed baseline and after 8th weeks. Measurement takes about 10 minutes.
  Static balance will be evaluated by the Y Balance Test.
Change on Dynamic Balance after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 10 minutes.
  Static balance will be evaluated by the Y Balance Test.
Change between baseline of Anaerobic Performance Tests-Vertical Jump Test and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 5 minutes.
  Vertical jump performance will be evaluated by the Counter Movement Jump.
Change between baseline of Anaerobic Performance Tests-Vertical Jump Test and after 8th week stretching exercise | Assessment will be performed baseline and after 8th weeks. Measurement takes about 5 minutes.
  Vertical jump performance will be evaluated by the Counter Movement Jump.
Change on Anaerobic Performance Tests-Vertical Jump Test and after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 5 minutes.
  Vertical jump performance will be evaluated by the Counter Movement Jump.
Change between baseline of Anaerobic Performance Tests-Horizontal Jump Test and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 5 minutes.
  Horizontal Jump Test will be used for horizontal evaluation of explosive force of lower extremities.
Change between baseline of Anaerobic Performance Tests-Horizontal Jump Test and after 8th week stretching exercise | Assessment will be performed baseline and after 8th weeks. Measurement takes about 5 minutes.
  Horizontal Jump Test will be used for horizontal evaluation of explosive force of lower extremities.
Change on Anaerobic Performance Tests-Horizontal Jump Test after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 5 minutes.
  Horizontal Jump Test will be used for horizontal evaluation of explosive force of lower extremities.
Change between baseline of Muscle Strength and after first stretching exercise | Assessment will be performed baseline and after first stretching. Measurement takes about 15 minutes.
  Muscle strength will be evaluated with isokinetic dynamometer in N /m.
Change between baseline of Muscle Strength and after 8th week stretching exercise | Assessment will be performed baseline and after 8th weeks. Measurement takes about 15 minutes.
  Muscle strength will be evaluated with isokinetic dynamometer in N /m.
Change on Muscle Strength after 6 week follow up period | The test will be performed after 6 weeks follow up period. It takes about 15 minutes.
  Muscle strength will be evaluated with isokinetic dynamometer in N /m.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Mani, MPT, Principal Investigator — Eastern Mediterranean University; Berkiye Kırmızıgil, DPT, Study Director — Eastern Mediterranean University; Emine H Tüzün, DPT, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Bouet V, Gahery Y. Muscular exercise improves knee position sense in humans. Neurosci Lett. 2000 Aug 4;289(2):143-6. doi: 10.1016/s0304-3940(00)01297-0. PMID 10904140
- [Background] Hassan BS, Mockett S, Doherty M. Static postural sway, proprioception, and maximal voluntary quadriceps contraction in patients with knee osteoarthritis and normal control subjects. Ann Rheum Dis. 2001 Jun;60(6):612-8. doi: 10.1136/ard.60.6.612. PMID 11350851
- [Background] Roijezon U, Clark NC, Treleaven J. Proprioception in musculoskeletal rehabilitation. Part 1: Basic science and principles of assessment and clinical interventions. Man Ther. 2015 Jun;20(3):368-77. doi: 10.1016/j.math.2015.01.008. Epub 2015 Jan 29. PMID 25703454
- [Background] Ghaffarinejad F, Taghizadeh S, Mohammadi F. Effect of static stretching of muscles surrounding the knee on knee joint position sense. Br J Sports Med. 2007 Oct;41(10):684-7. doi: 10.1136/bjsm.2006.032425. Epub 2007 May 17. PMID 17510229
- [Background] Bjorklund M, Hamberg J, Crenshaw AG. Sensory adaptation after a 2-week stretching regimen of the rectus femoris muscle. Arch Phys Med Rehabil. 2001 Sep;82(9):1245-50. doi: 10.1053/apmr.2001.24224. PMID 11552198
- [Background] Larsen R, Lund H, Christensen R, Rogind H, Danneskiold-Samsoe B, Bliddal H. Effect of static stretching of quadriceps and hamstring muscles on knee joint position sense. Br J Sports Med. 2005 Jan;39(1):43-6. doi: 10.1136/bjsm.2003.011056. PMID 15618341
- [Background] Streepey JW, Mock MJ, Riskowski JL, Vanwye WR, Vitvitskiy BM, Mikesky AE. Effects of quadriceps and hamstrings proprioceptive neuromuscular facilitation stretching on knee movement sensation. J Strength Cond Res. 2010 Apr;24(4):1037-42. doi: 10.1519/JSC.0b013e3181d09e87. PMID 20300021
- [Background] Pincivero DM, Bachmeier B, Coelho AJ. The effects of joint angle and reliability on knee proprioception. Med Sci Sports Exerc. 2001 Oct;33(10):1708-12. doi: 10.1097/00005768-200110000-00015. PMID 11581556
- [Derived] Mani E, Kirmizigil B, Tuzun EH. Effects of two different stretching techniques on proprioception and hamstring flexibility: a pilot study. J Comp Eff Res. 2021 Sep;10(13):987-999. doi: 10.2217/cer-2021-0040. Epub 2021 Jul 7. PMID 34231374